CLINICAL TRIAL: NCT05668247
Title: The Effects on Sleep Quality and Fatıgue Level of Foot Bath Made in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Effects on Sleep qualıty and fatıgue Level of Foot Bath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevil Şahin (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Sevil Şahin, Associate Professor, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/370
Record Dates: First submitted 2022-12-09; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; fatigue; foot bath; nursing; sleep quality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): foot bath is a type of relaxation and care performed by putting feet in water. Feet, as the organs carrying the whole body weight are the body parts where fatigue is felt most. In this study, a specially designed foot bath bucket was used in order to apply foot bath for the patients in the experimental group. The bucket has a five-level water heating system (35-48 °C). It has a magnetic field and operates at 390 Watt. It has a splash shield. There are non-slip rubber legs on its bottom. it has heat protection feature for thermal insulation as it has a two-walled structure
  Interventions: Other: FOOT BATH
- Control (No Intervention): On the first day (the first follow-up), Patient Information Form, PSQI (ANNEX-II) and Piper Fatigue Scale were applied to the patients in the control group whose consent was obtained in the first follow-up, through face-to-face interview. At the end of the 30th day (the second follow-up), PSQI and Piper Fatigue Scale were applied again to the patients who came for the outpatient clinic control.
  The routine treatment of the control group was not interfered and no intervention was performed.

INTERVENTIONS:
Other: FOOT BATH — In general, foot bath is a type of relaxation and care performed by putting feet in water. Feet, as the organs carrying the whole body weight are the body parts where fatigue is felt most. In this study, a specially designed foot bath bucket was used in order to apply foot bath for the patients in the experimental group.
  Arms: Intervention

SUMMARY:
Aims and objectives: To determine the effect of foot bath on sleep quality and fatigue level in patients with chronic obstructive pulmonary disease (COPD).

Background: İnsomnia and fatigue are one of the most common symptoms in people with COPD and adversely affects their activities of daily living.

Design: This study was conducted as a nonrandomized controlled trial. Methods:The study sample comprised 70 patients who met the inclusion criteria.Data were collected with Patient Information Form, Pittsburgh Sleep Quality Index and Piper Fatigue Scale. Intervention group; The 30-day foot bath was administered for 10 minutes before bedtime, while no control was performed in the control group. The Pittsburgh Sleep Quality Index (PUKI) and the Piper Fatigue Scale were administered in both groups at the beginning of the service (first follow-up) and four weeks later (second follow-up) at the outpatient clinic.

Conclusions: The foot bath by individuals with COPD was determined to significantly improve the participants'levels sleep quality and fatigue.

DETAILED DESCRIPTION:
The physical symptoms frequently seen in COPD patients and adversely affecting routine life are dyspnoea, cough, phlegm, malnourishment/loss of appetite, nausea-vomiting, constipation, dehydration, sleeplessness, weakness/fatigue, delirium, anxiety, and depression.

It has been stated that the patients who experience severe symptoms cannot sleep, this condition impairs their sleep quality and they feel fatigue all day long. It has been observed in the literature that there are a decrease in sleep efficiency and total sleep duration, an increase in sleep latency, falling asleep late, and waking up, and a decrease in non-rapid eye movement (NREM) sleep and rapid eye movement (REM) sleep among COPD patients especially due to the cough and respiratory distress symptoms.

1.2 Literature review The qualitative aspects of sleep include sleep duration, sleep latency and the number of awakening during the night; on the other hand, its subjective aspects include elements such as sleep depth and relaxation. It is important to assess these elements in order to assess the sleep quality of patients.

Just like the sleep problems, fatigue is also an important problem seen in patients with COPD. In the studies, it has been determined that the patients with COPD have different levels of fatigue and their mental, physical and social functions may be affected from fatigue.

It is thought that the most common symptom in patients with chronic obstructive pulmonary disease (COPD) is dyspnoea. However, it has been reported that fatigue is observed in the patients as frequent as respiratory distress. Fatigue is the main factor restricting the exercise tolerance of the individuals. A positive significant correlation has been determined between fatigue and dyspnoea. Fatigue affects the realisation of activities of daily living negatively and impairs quality of life as it reduces activity tolerance of patients.

Decreased effect of the pharmacological methods mostly preferred to solve sleep problems, the side effects of drugs, and the necessity of using drugs continuously have led people to use non-pharmacological methods. These methods include the complementary and integrative practices such as yoga, aromatherapy, massage, energy therapy, music therapy, reflexology, acupuncture, and acupressure. In recent years, many complementary and integrative methods have come into use as the number of studies on eliminating sleep problems and enhancing sleep quality has increased. One of these methods is hot foot bath. It is stated that hot foot bath provides a relaxing body temperature by regulating blood circulation, keeping feet in hot water relaxes the whole body, reduces fatigue and makes sleeping easier and, therefore, it is a therapeutic technique frequently used in nursing.

Important tasks of nurses include preparing the suitable environment for the patients to take a rest and providing to fulfil the basic physiological needs such as sleep etc. to enable the human body to continue its existence. For this reason, determining the factors preventing the patients from sleeping well in the hospital environment and eliminating these factors are of prime importance. Nurses who are the members of the healthcare team should solve the problems caused by sleeplessness and prevent the fatigue problem that may be caused by sleeplessness.

This study was conducted to examine the effect of the hot foot bath on sleep quality and fatigue level of the individuals with COPD.

The hypotheses of the study were as follows:

H1: The foot bath applied with hot water at 38-40°C for 10 minutes before going to sleep for 30 days is effective in enhancing sleep quality of the individuals staying in the hospital and receiving COPD treatment.

H2: The foot bath applied with hot water at 38-40°C for 10 minutes before going to sleep for 30 days is effective in decreasing fatigue level of the individuals staying in the hospital and receiving COPD treatment.

ELIGIBILITY:
Inclusion Criteria:

The patients,

* who were diagnosed with COPD,
* were aged between 55-85 years,
* did not have a psychiatric disease requiring treatment,
* had no diagnosed sleep disorder,
* had orientation to person, place, and time, can be communicated verbally,
* had a general state of health enough to perceive the questions in the questionnaire and answer them correctly,
* had a mild (FEV1 ≥ 80%) and moderate (50% ≤ FEV1 < 80%) COPD stage,
* agreed to participate in the study were included in the study.

Exclusion Criteria:

The patients,

* who had Diabetes Mellitus (DM), CVA, CHF, coronary artery disease, coagulation disorders such as varicosity, deep vein thrombosis and disseminated intravascular coagulation,
* were using CPAP (Continuous Positive Airway Pressure) and BIPAP (Bi-level Positive Airway Pressure) devices,
* were diagnosed with sleep disorder,
* had the general condition disorder developed related to diagnosis within the application and control process were excluded from the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Hypotes 1 | Ahrough study completion, an average of 1 year
  The foot bath applied with hot water at 38-40°C for 10 minutes before going to sleep for 30 days is effective in enhancing sleep quality of the individuals staying in the hospital and receiving COPD treatment.
Hypotes 2 | hrough study completion, an average of 1 year
  The foot bath applied with hot water at 38-40°C for 10 minutes before going to sleep for 30 days is effective in decreasing fatigue level of the individuals staying in the hospital and receiving COPD treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sevil Şahin, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No